CLINICAL TRIAL: NCT06194006
Title: Long-term Follow-up of Huntington's Disease Patients Treated With Intrastriatal Fetal Neuron Allograft
Brief Title: Long Term Follow-up Grafted Huntington's Disease Patients
Acronym: Post-MIGHD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K140601J; 2018-A02569-46 (Other: IDRCB)
Record Dates: First submitted 2022-03-09; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-05

CONDITIONS: Huntington Disease
Keywords: Grafted patients; Long term follow-up
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long term follow-up (Other): * Formalized and standardized follow-up
  * Retrospective data collection
  * Biological collections
  * Biological collections's centralisation
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Follow-up grafted patients as long as their condition allows

SUMMARY:
Long-term follow-up of Huntington's disease patients treated with intrastriatal allografts is essential to assess the benefit/risk ratio of grafts as well as their effectiveness. Indeed, some patients are likely to develop adverse effects and the impact of alloimmunisation phenomena remains to be explored.

DETAILED DESCRIPTION:
The aim is to create a specific cohort of transplant patients, to homogenise their follow-up methods, to collect all the patient data (medical, paramedical, imaging, biological) acquired from the end of their participation in MIG-HD'study (Foetal Striatal allografting in Huntington's disease: a multicentre, randomised, delayed start, phase 2 open-label cell therapy trial) until the last possible follow-up of the last patient in the study

ELIGIBILITY:
Inclusion Criteria:

* Adult patients transplanted under the MIG-HD protocol
* Information and informed consent from patients or their representative
* Affiliation with a social security scheme or beneficiary

Exclusion Criteria:

* Patient under AME
* Patient unable to express consent and not subject to legal protection
* Knowned pregnancy or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2034-01-01 (Estimated); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression of the Unified Huntington's Disease Rating Scale (UHDRS) motor score | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Progression of the Unified Huntington's Disease Rating Scale For Advanced Patients (UHDRS-FAP) motor score | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient

SECONDARY OUTCOMES:
Slopes comparison of neurological scores (Unified Huntington's Disease Rating Scale (UHDRS) or Unified Huntington's Disease Rating Scale For Advanced Patients (UHDRS-FAP)) before and after transplantation | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Slopes comparison of cognitive scores (Unified Huntington's Disease Rating Scale (UHDRS) or Unified Huntington's Disease Rating Scale For Advanced Patients (UHDRS-FAP)) before and after transplantation | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Slopes comparison of psychiatric scores (Unified Huntington's Disease Rating Scale (UHDRS) or Unified Huntington's Disease Rating Scale For Advanced Patients (UHDRS-FAP)) before and after transplantation | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Slopes comparison of neuropsychologic scores (Mattis Dementia Rating Scale/Trail Making test/Hopkins Verbal Learning Test/Categorical fluency/Sign barrier test/Montgomery-Åsberg Depression Rating Scale (MADRS)) before and after transplantation | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Comparison of the clinical evolution (Unified Huntington's Disease Rating Scale (UHDRS) or Unified Huntington's Disease Rating Scale For Advanced Patients (UHDRS-FAP)) of transplanted patients with that of non-transplanted patients in the BioHD cohort | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  Grafted patients and cohort patients (BIOHD)
Events and adverse reactions recording since the transplantation | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Research and identification of anti-MHC Ab from samples acquired under the MIG-HD and Post-MIGHD protocols as well as in care | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Correlation between graft activity measured by imaging and patient performance | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Correlation between post-mortem observations of the brains of deceased patients and measurements obtained by MRI and PET-SCAN in studies MIG-HD and BioHD | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Correlation between post-mortem brain observations and patient performance before death | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient
Analysis of brains collected as part of MIG-HD and POST-MIGHD i) to quantify neuropathological lesions ii) to search for markers of inflammatory reactions | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For all patients whose brains have been recovered
Research into predictive factors (relationships between fetal haplotypes, patient haplotypes and appearance of alloimmunization phenomena) of the evolution of transplanted patients | From the end of participation at MIGHD's study until the death from any cause or assessed up to 10 years after consentement signed
  For each patient

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Catherine BACHOUD-LEVI, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - Hôpital Henri Mondor, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWNED BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION